CLINICAL TRIAL: NCT06851273
Title: National Implementation of Highly Efficient Evidence-Informed Treatment for Youth with Eating Disorders
Brief Title: Guided Self Help for Eating Disorders Implementation Study
Acronym: GSHimplement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jennifer Couturier, Principal Investigator, McMaster University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 18545
Record Dates: First submitted 2025-02-12; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Eating Disorders
Keywords: Anorexia nervosa; Mental disorders; Adolescent eating disorders; Psychotherapy intervention; Guided self help therapy; Family-based treatment
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Parents who have a child with anorexia nervosa (Experimental): Each participant will receive a series of pre-recorded videos, an electric scale, and a therapy manual ("Help Your Teen Beat an Eating Disorder"). This will include content on empowering parents to renourish their child and interrupt binge/purge behaviors.
  Interventions: Behavioral: Guided Self Help Family Based Therapy (GSH FBT)

INTERVENTIONS:
Behavioral: Guided Self Help Family Based Therapy (GSH FBT) — Each family will participate in ten virtual sessions of GSH FBT with a trained GSH practitioner local to their provincial study site. Parents will meet their coach for a 60-minute onboarding session where the parents/caregivers are familiarized with the video platform used in treatment. Then, the treatment consists of ten virtual 20-minute sessions over 6 months. In GSH FBT, the parents weigh the adolescent patient prior to the session, on the same day as the session, and report the weight to the coach. Throughout treatment, parents have access to an online platform with a series of videos that outline the core components of FBT: the urgency to act, parental empowerment, medical complications, strategies to use during and after mealtime, and how to externalize the illness. In line with GSH approaches, coach-therapists direct parents to watch or review videos and text content rather than directly affecting behavioral change.

SUMMARY:
Eating disorders are amongst the most understudied illnesses affecting young women in Canada. Further, mortality rates are amongst the highest of all psychiatric illnesses. Despite their high prevalence and mortality rates, research into adolescent eating disorders is underfunded in Canada. In addition to the problem of research underfunding, healthcare system underfunding exists - creating long waiting lists and fragmented care for children and youth with eating disorders. More efficient treatments are urgently needed to reduce wait times and provide expedited care to adolescents on eating disorder waitlists. The current study aims to assess whether implementing a virtual parent-lead therapy, Guided Self Help Family-Based Therapy (GSH FBT) might alleviate wait times for eating disorder services and also reduce eating disorder symptomatology in young people with anorexia nervosa. This study also aims to determine the experiences of both families and medical teams of GSH FBT implementation as an intervention.

DETAILED DESCRIPTION:
The most widely used evidence-based treatment for children and adolescents with eating disorders is Family-Based Treatment (FBT). Similarly, Guided Self-Help FBT (GSH FBT) is a virtual treatment, adapted using FBT principles, that involves a therapist "coach" and a video platform for parents. Therapeutic challenges such as treatment fidelity could be partially mitigated with a model, such as GSH FBT, in which essential material is delivered by video or written material, standardizing the treatment and ensuring that key components are delivered. Given the surging wait list times for adolescent eating disorder treatment, GSH FBT is emerging as a promising, more efficient alternative to longer-term FBT and FBT-V. This study is aimed at examining the implementation of GSH FBT for pediatric patients with eating disorders across nine provinces in Canada using a mixed methods design. To implement this new model of care, the investigators will use implementation teams at each site along with GSH FBT provider training and consultation. The investigators will evaluate the implementation approach using qualitative and quantitative methods including fidelity assessments, examination of wait times, patient, family, and provider outcomes, as well as the overall experience of the implementation of the intervention. Experience of implementation will be assessed using qualitative measures such as semi-structured interviews and focus groups.

ELIGIBILITY:
Inclusion Criteria:

* Family including an adolescent with a confirmed diagnosis of Anorexia nervosa according to DSM-5-TR criteria.
* Access to computer and internet connection
* Have the capacity to speak, write, and understand English
* Therapist/coaches are licensed mental health clinician with experience in eating disorder treatment

Exclusion Criteria:

* Adolescent has a current physical or mental disorder that requires hospitalization and/or prohibits the use of psychotherapy
* Adolescent has a current dependence on drugs or alcohol
* Adolescent has a current physical condition known to influence weight or eating (pregnancy, diabetes mellitus)
* Adolescent has expected body weight of less than 75%
* Adolescent/family has undergone four or more sessions of FBT for anorexia nervosa at any time
* Does not have the capacity to speak, write, and understand English
* Does not have access to computer and internet connection
* Professionals are not licensed mental health professionals with experience in eating disorder treatment.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Implementation success at participating sites, as measured by fidelity to GSH FBT model | Immediately after each session throughout the 10-week protocol
  Fidelity of therapists will be measured via administration of a self-reporting fidelity questionnaire piloted in a previous GSH FBT feasibility study. This questionnaire includes nine yes/no questions that gauge whether the therapist was adherent to GSH FBT principles: 1) ensuring only parents are present; 2) ensuring the adolescent is not present; 3) asking parents questions/comments about course materials; 4) avoiding direct orchestration of behavioural change; 5) referencing course materials during the session; 6) focusing the session on treatment; 7) assigning homework appropriately; and 8) & 9) verifying session length. Videos will also be monitored regularly for fidelity via expert review.

SECONDARY OUTCOMES:
Changes in wait times as result of implementation approach | at the baseline (week 0) and at the end of treatment (24 weeks)
  Changes in wait time for service will be assessed by asking site administrators to provide wait time for service (in days) and an estimate of number of adolescents waiting for eating disorder services.
Changes in severity of eating disorder symptoms | at the baseline (week 0) and at the end of treatment (24 weeks)
  Changes in severity of eating disorder symptoms will be assessed using the Eating Disorder Examination Questionnaire (EDEQ), a 28-item standardized questionnaire that measures the severity of symptoms of eating disorders. The EDEQ is scored using a 7-point, forced-choice rating scale (0-6) with scores of 4 or higher indicative of clinical range and severity of the illness.
Changes in severity of depressive symptoms | at the baseline (week 0) and at the end of treatment (24 weeks)
  Changes in severity of depressive symptoms will be assessed using the Beck Depression Inventory (BDI), a 21-item questionnaire used to measure the severity of depressive symptoms. Minimum score is 0, maximum score is 63.
Changes in anxiety symptoms | at the baseline (week 0) and at the end of treatment (24 weeks)
  Changes in severity of anxiety symptoms will be assessed using the Beck Anxiety Inventory (BAI), a 21-item questionnaire used to measure the severity of anxiety symptoms. Minimum score is 0, maximum score is 63.
Changes in obsessional thinking and compulsive behaviours (linked to eating disorder symptomatology) | at the baseline (week 0) and at the end of treatment (24 weeks)
  Changes in severity of obsessional thinking and compulsive behaviours (linked to eating disorder symptomatology) will be assessed using the Yale-Brown-Cornell Eating Disorder Scale (YBC-EDS), It includes a comprehensive checklist of 21 preoccupations and 44 rituals related to food, eating, weight, shape, and appearance. Each item is rated on a scale from 0 to 4, with 0 indicating no symptoms and 4 indicating very severe symptoms. The total score is the sum of these individual ratings. Therefore, the minimum possible score is 0 (indicating no symptoms), and the maximum possible score is 260 (indicating the most severe symptoms).
Changes in obsessional thinking and compulsive behaviours | at the baseline (week 0) and at the end of treatment (24 weeks)
  Changes in severity of obsessional thinking and compulsive behaviours will be assessed using the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS-II), a self-report questionnaire assessing obsessions and compulsions separately from eating disorder symptomatology, will also be used to assess this outcome. The total score ranges from 0 (least severe) to 50 (most severe).
Changes in parental self-efficacy | at the baseline (week 0) and at the end of treatment (24 weeks)
  Changes in parental self-efficacy will be assessed using the "Parents versus Eating Disorder Scale" (PvED), a 7-item measure assessing parental self-efficacy related to re-feeding their child with an eating disorder. Scores range from 7 (least severe) to 35 (most severe).
Provider's readiness for change | at the baseline (week 0) and at the end of treatment (24 weeks)
  Provider individual readiness for change will be evaluated using the Brief Individual Readiness for Change Scale (BIRCS), administered to therapist-coaches. Minimum score is 0, maximum score is 20.
Providers' attitudes towards evidence-based practice | at the baseline (week 0) and at the end of treatment (24 weeks)
  Provider attitudes about evidence-based practice will be assessed using the Evidence Based Practice Attitudes Scale (EBPAS), administered to therapist-coaches. Minimum score for each subscale is 0, maximum score for each subscale is 4.
Provider's confidence in ability to deliver intervention | at the baseline (week 0) and at the end of treatment (24 weeks)
  Confidence related to the intervention will be assessed by administering an adapted version of the Perceived Attributes of the Principles of Effectiveness Scale (MPAQ) to therapist-coaches. The minimum score is 18, the maximum score is 90.

OTHER OUTCOMES:
The experience of parents/families participating in GSH FBT treatment | Interviews with families will be scheduled within two weeks of their provider notifying us that their final treatment session has occurred.
  Experiences of families participating in GSH FBT treatment will be qualitatively measured by semi-structured interviews with each family.
Implementation teams' experiences of GSH FBT treatment and its implementation | Focus groups with a site will occur within two weeks of when the investigators have been notified that all GSH FBT sessions have been completed at the site.
  Implementation teams' experiences of GSH FBT treatment and implementation will be qualitatively measured by semi-structured focus groups with each site team.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Couturier J, Smith J, Nicula M, Nella E, Yanover T, Agostino H, Annema S, Boman J, Bond J, Coelho JS, Coolen AM, Datta N, Dimitropoulos G, Ford C, Isserlin L, Johnson N, Jones S, Katzman D, Kelly B, Keshen A, Kimber M, Kumar S, Kurji A, Lacroix E, Markland A, Matheson B, McVey G, McQuillan B, Norris M, Obeid N, Phillips S, Preskow W, Rodrigues A, Smith S, Soroka C, Spettigue W, Webb C, Wournell J, Lock JD. National implementation of guided self-help family-based treatment for youth with eating disorders: a study protocol. BMC Psychiatry. 2025 Nov 6;25(1):1066. doi: 10.1186/s12888-025-07545-1. PMID 41199206